CLINICAL TRIAL: NCT05106556
Title: The Effect of Respiratory Muscle Training on Respiratory Parameters, Functional Capacity, Balance and Quality of Life in Interstitial Lung Patients
Brief Title: Effect of Respiratory Muscle Training in Interstitial Lung Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Onur Aydın, Lecturer, PT, PhD (c), Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BezmialemVU-AYDIN-001
Record Dates: First submitted 2021-10-13; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Interstitial Lung Disease
Keywords: Interstitial lung disease; Interstitial pulmonary fibrosis; Sarcoidosis; Respiratory muscle training; Pulmonary Function; Functional Capacity; Physiotherapy; Balance; Quality of Life; 6 Minute Walk Test
MeSH Terms: conditions — Lung Diseases, Interstitial; Pulmonary Fibrosis; Sarcoidosis

STUDY DESIGN:
Intervention Model Description: Group 1: Inspiratory Muscle Training (IMT) Group Group 2: Control Group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive conventional chest physiotherapy, two times a day, 5 days a week for 8 weeks. After the training given by the physiotherapist one exercise session will be supervised in a clinic per week, other sessions will be performed at home.
  Maximal inspiratory mouth pressure measurements will be measured once a week to eliminate the effect of learning, however the training intensity will remain at the lowest intensity of the device for 8 weeks and will not be increased.
  Interventions: Other: Conventional Chest Physiotherapy
- Inspiratory Muscle Training (IMT) Group (Experimental): In addition to conventional chest physiotherapy programme, patients in this group will also receive inspiratory muscle training at %30 of the maximal inspiratory mouth pressure (MIP) value of at least five days a week, for 15 minutes twice days, for 8 weeks at home. One exercise session will be supervised in a clinic per week, other sessions will be performed at home.
  Maximal inspiratory mouth pressure measurements will be measured once a week. The training intensity will be increased weekly. At this rate it is 30% of the maximal inspiratory pressure value.
  Interventions: Other: Conventional Chest Physiotherapy; Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Conventional Chest Physiotherapy — Programme will include diaphragmatic breathing exercise, pursed lip breathing exercise, thoracic expansion exercises, upper and lower extremity exercises, stretching the pectoral muscles, posture exercises, walking training and teaching respiratory control.
Other: Inspiratory Muscle Training — Threshold IMT device will be used for the training. Training intensity will set at 30% of the maximum inspiratory pressure with the threshold loading method.
  Arms: Inspiratory Muscle Training (IMT) Group

SUMMARY:
The aim of this study is to investigate the possible effects of inspiratory muscle training (IMT) on respiratory functions, functional capacity, balance and quality of life in patients with interstitial lung disease.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) include a heterogeneous group of progressive, acute and chronic diseases that diffusely affect the lung and characterized by varying degrees of inflammation and fibrosis in the lung parenchyma. The disease group usually shows a restrictive pattern and progresses with gas exchange abnormalities.

Progressive lung fibrosis was first described in 1935. Over the years, more than 150 lung disease characterized by acute or chronic pulmonary fibrosis of varying degrees with known or unknown cause have been defined and these diseases were named interstitial lung disease (ILD) in 1970s. Common symptoms in chronic interstitial lung diseases in general; dyspnea, dry cough, exercise intolerance and fatigue. All these features of interstitial lung diseases cause an increase in respiratory work and ventilatory deterioration in exercise. Apart from these general features, muscle weakness and related exercise intolerance may occur in some specific conditions.

The most important factor limiting exercise capacity in these patients is circulatory disorder, which cause exercise induced deterioration in gas exchange. Hypoxemia induced exercise intolerance causes a decrease in health-related quality of life, limitation of functional capacity and inactivity in daily life.

According to the American Thoracic Society (ATS) / European Respiratory Society (ERS) respiratory rehabilitation guideline, although the data are not conclusive, inspiratory muscle training is recommended as an adjunct to pulmonary rehabilitation, especially in patients with suspected or confirmed respiratory muscle weakness. The effect of well-structured and supervised inspiratory muscle training (IMT) on respiratory functions, diaphragm weakness, functional capacity, balance and quality of life in patients with interstitial lung disease is unknown.

It is important that this research will be carried out in this area and because it has a current subject.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with interstitial lung disease (idiopathic pulmonary fibrosis, collagen vascular diseases, sarcoidosis, etc.),
* Being clinically stable,
* Not receiving supplemental oxygen therapy,
* No pulmonary infection in the last 6 weeks,
* Being ambulation.

Exclusion Criteria:

* Presence of obstructive pulmonary disease such as chronic obstructive pulmonary disease (COPD), asthma, bronchiectasis
* Presence of a history of effort-induced syncope
* Presence of severe orthopedic or neurological disease
* Presence of unstable serious cardiac disease

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-01-03 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Respiratory Function Test / Forced Vital Capacity (FVC) | Eight weeks
  Change from baseline Forced Vital Capacity (FVC) in respiratory function test at 8 weeks. FVC will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Respiratory Function Test / Forced Expiratory Volume 1 second (FEV1) | Eight weeks
  Change from baseline Forced Expiratory Volume 1 second (FEV1) in respiratory function test at 8 weeks. FEV1 will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Respiratory Function Test / Peak Expiratory Flow (PEF) | Eight weeks
  Change from baseline Peak Expiratory Flow (PEF) in respiratory function test at 8 weeks. PEF will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Respiratory Function Test / Tiffeneau-Pinelli index (FEV1/FVC) | Eight weeks
  Change from baseline Tiffeneau-Pinelli index (Forced Expiratory Volume 1 second (FEV1) / Forced Vital Capacity (FVC)) in respiratory function test at 8 weeks. FEV1 / FVC will be evaluated using spirometry, according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Respiratory Muscle Strength / Maximum Inspiratory Pressure (MIP) | Eight weeks
  Change from baseline Maximum Inspiratory Pressure (MIP) at 8 weeks. Respiratory muscle strength will be measured according to the portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical UK), American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Respiratory Muscle Strength / Maximum Expiratory Pressure (MEP) | Eight weeks
  Change from baseline Maximum Expiratory Pressure (MEP) at 8 weeks. Respiratory muscle strength will be measured according to the portable, electronic intraoral pressure measuring device (MicroRPM, Micro Medical UK), American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Functional Capacity | Eight weeks
  Change from baseline distance covered in six-minute walk test at 8 weeks
Balance / Postural Stability | Eight weeks
  Change from baseline postural stability test score in Biodex Balance System at 8 weeks
Balance / Limits of Stability | Eight weeks
  Change from baseline limits of stability test score in Biodex Balance System SD at 8 weeks
Balance / Sensory Integration and Balance Test Score | Eight weeks
  Change from baseline sensory integration and balance test score in Biodex Balance System SD at 8 weeks

SECONDARY OUTCOMES:
Peripheral Muscle Strength | Eight weeks
  Change from baseline M. Quadriceps strength at 8 weeks. It will be performed using an electronic hand dynamometer (Commander Muscle Tester; JTECH Medical, USA). M. Quadriceps muscle strength will be measured; it will evaluate the isometric muscle strength of that muscle by applying maximum resistance to the M. Quadriceps muscle with the electronic hand dynamometer.
Pain Level | Eight weeks
  Change from baseline Visual Analogue Scale (VAS) at 8 weeks.This scale consists of a horizontal, straight line. The line has a value of 0 at the beginning and a value of 10 at the end. A value of 0 means no pain, a value of 10 means unbearable pain. high values represent severe pain.
Dyspnea | Eight weeks
  Change from baseline Modified Medical Research Council Dyspnea Scale (mMRC) at 8 weeks. The Modified Medical Research Council Dyspnea Scale (mMRC) is a five-item scale based on various activities that cause breathlessness. The scale is rated from "0" to "4". High values indicate severe shortness of breath.
Health-Related Quality of Life | Eight weeks
  Change from baseline St. George's Respiratory Questionnaire (SGRQ) at 8 weeks. St. George's Respiratory Questionnaire consists of 76 questions that can be filled in about 15 minutes. It consists of 3 subgroups that evaluate respiratory symptoms (dyspnea, cough, sputum, wheezing, severity and frequency), activity status (physical functions that cause shortness of breath, housework, hobbies) and the impact of the disease (social activities and psychological state). The three parts of the test are scored separately and the total score is calculated. Scores range from 0-100. A score of zero indicates normal and a score of 100 indicates maximum disability.

CONTACTS AND LOCATIONS:
Overall Officials: Onur AYDIN, PhD (c), Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih/Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No